CLINICAL TRIAL: NCT01031238
Title: Pilot Study to Compare the PEM Uptake Value (PUV) and Standardized Uptake Value (SUV) in Patients With Malignancies of the Breast
Brief Title: Comparison of PEM Uptake Value (PUV) and Standardized Uptake Value (SUV) in Patients With Malignancies of the Breast
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-0479
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer
Keywords: PEM Uptake Value; PUV; Standardized Uptake Value; SUV; Malignancies of the Breast; [18F]-FDG-PET/CT scanning; Tumor; positron emission tomography/computed tomography; PET/CT scan
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this clinical research study is to learn if using the PEMFlex Solo II, a high-resolution camera for positron emission tomography (PET) scan imaging, on an area of the body that has, or is suspected to have cancer will give researchers the same or better information about the disease compared to the images taken with a routine PET/computed tomography (CT).

Researchers will compare the images taken using the PEMFlex Solo II to the images taken during your scheduled routine PET/CT scan, as well as any additional routine CT scan(s), magnetic resonance imaging (MRI) scan(s), and/or ultrasound image(s) you may have had within the last 30 days or may have in the next 30 days.

DETAILED DESCRIPTION:
If you agree to take part in this study, right after your already scheduled routine PET/CT scan is complete, a study staff member will take you to a separate imaging room located in the same clinic area where your routine PET/CT scan was just performed.

You will then sit in a chair as a study staff member positions the PEMFlex Solo II on either side of your breast that has, or is suspected to have cancer. To take images using the PEMFlex Solo II, the breast is placed between two flat panels on the scanning machine and compressed (flattened). The position of the breast for this procedure is similar to getting a mammogram, but the PEMFlex Solo II uses about 50% less force to compress the breast(s). The compression will be repeated on the other breast if you are having scans of both breasts performed.

It will take about 20 minutes to set up the PEMFlex Solo II and take the PET scan images.

Length of Study:

After the PET scan images have been taken using the PEMFlex Solo II, your participation in this study will be over.

This is an investigational study. The PEMFlex Solo II is commercially available for PET scan imaging of the breast.

Up to 24 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. A signed informed consent.
2. Known or suspected malignancy involving the breast as determined by biopsy, physical examination or noninvasive imaging studies including plain films, CT, MR, ultrasound or nuclear medicine imaging.
3. Scheduled for routine clinical imaging at the ACB PET/CT facility.
4. Participant must be at least 18 years of age.

Exclusion Criteria:

1. Uncontrolled blood glucose levels (>200 mg/dl).
2. Patient is unable to comprehend the requirements of the study.
3. Patient is unable to undergo scanning of the known or suspected lesion with the high-resolution PEM (PET) scanner (due to body habitus, inability to comply with positioning requirements, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known or suspected tumors of the breast, 18 years or older scheduled for routine clinical imaging at the PET/CT facility.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2009-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Correlation between PUV and SUV of breast malignancies in patients undergoing [18F]-FDG-PET/CT scanning | 20 minutes for imaging using PEMFlex Solo II
  Formal quantitative assessment of the correlation between PUVmax values and maximum standardized uptake value (SUVmax) values performed by testing whether the Pearson correlation between these values exceeds 0.7.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Rohren, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org